CLINICAL TRIAL: NCT05523388
Title: RoLSSroice - Role of Spinal Load in the Pathophysiology of Lumbar Spinal Stenosis: A Translational Approach Combining Clinical and Radiological Parameters, in Vivo Biomechanical Experiments and Advanced in Silico Musculoskeletal Modeling
Brief Title: Role of Spinal Load in the Pathophysiology of Lumbar Spinal Stenosis
Acronym: RoLSSroice
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01170; mu22Netzer3
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Spinal Stenosis
Keywords: patient-reported outcome measures (PROMs); symptomatic lumbar spinal stenosis sLSS); Oswestry disability index (ODI); postural biomechanical analysis; ambulatory biomechanical analysis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collection of health-related data — A multimodal set of data including experimental, clinical, functional, radiological and biomechanical data is compiled before and after routine surgical intervention at baseline and at one-year follow-up.

SUMMARY:
This study is to improve the understanding of the role of postural and ambulatory biomechanics for symptoms in patients with sLSS and to correlate patient-reported outcome measures (PROMs) with dynamic compensation (difference between static and dynamic sagittal spinal alignment) in patients with symptomatic lumbar spinal stenosis sLSS).

DETAILED DESCRIPTION:
Lumbar spinal stenosis (LSS) is a common syndrome affecting the human spine characterized by age related degeneration of the lumbar discs, facet joints (FJs) and hypertrophy of the ligamentum flavum resulting in pain, limited function and compromised quality of life. Understanding the interrelationship between spinal load, kinematics and functional disability is one of the key factors in the prevention of this disease. This project assesses sagittal spinal balance and motion in patients with sLSS using an optoelectronic method based on infrared cameras and retroreflective markers and elicits paraspinal muscle fatigue using a modified version of the Biering-Sørensen test and compares sagittal spinal balance and motion before and after the fatigue exercise, which will allow to associate sLSS-specific motion patterns to paraspinal muscle fatigue. Additional data generated using magnetic resonance imaging (MRI) allows detecting associations between sLSS, muscle degeneration and fatty infiltration. Radiological images from the spine will be obtained in upright position using EOS®, a specialized low-dose x-ray unit. These images will allow the calculation of the anatomical global and local sagittal spinal balance, enabling a characterization of spinal kinematics in patients with sLSS and a validation of the workflow based on the optoelectronic method. Coded data obtained from EOS and motion analysis will allow optimizing existing biomechanical musculoskeletal models of the human spine. The results of this study will provide first mechanistic evidence of the role of clinical, radiological, functional and biomechanical factors in spine load. The combination of in vivo experiments with in silico experiments represents a unique opportunity of translating knowledge gained from systematic experiments considering biological measurements back to the patient. This study is to improve the understanding of the role of postural and ambulatory biomechanics for symptoms in patients with sLSS.

ELIGIBILITY:
Inclusion Criteria:

* age > 30 years
* BMI < 35 kg/m2
* diagnosed sLSS
* clinical symptoms for at least 6 months
* intermittent neurogenic claudication with limitations of their walking ability due to symptoms in the lower back and or in one or both legs
* unsuccessful conservative treatment
* confirmation of the LSS through MRI
* scheduled for surgery

Exclusion Criteria:

* inability to provide informed consent
* previous spine surgery
* use of walking aids
* other neurologic disorders affecting gait
* MRI incompatibility
* pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Department of Spine Surgery at the University Hospital Basel. The surgical procedure is not affected by the study and is not subject of investigation.
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry disability index (ODI) | At baseline and at one-year follow-up
  Disability related to sLSS will be assessed with the ODI, which is considered the gold standard of low back functional outcome tools. The ODI is a questionnaire comprising 10 self-administered items that quantify a patient's perceived level of functional disability. Each of the items relates to a different area of functional impairment and consists of six statements, which are scored from zero to five points.
Change in Dynamic compensation | At baseline and at one-year follow-up
  Dynamic compensation is defined as the difference between static and dynamic sagittal spinal alignment. Six possible gait events are available to choose from for the definition of dynamic sagittal spinal balance (left and right; heel-strike, toe-off, midstance). Dynamic sagittal spinal balance may be defined as sagittal spinal balance during left/right midstance, left/right heel strike and/or left/right toe off. The most appropriate gait event to calculate dynamic sagittal spinal balance will be used.

SECONDARY OUTCOMES:
Change in Sagittal spinal balance assessed using motion capture | At baseline and at one-year follow-up
  The curvature of the lumbar and thoracic spine during stance and during walking will be computed from the marker data using MATLAB™ software. A cubic polynomial function will be fitted to the marker positions in each time frame, approximating an S-shaped spine curvature with thoracic kyphosis (TK) and lumbar lordosis (LL) curves. The workflow used to calculate sagittal spinal balance parameters is based on the calculation methods for radiological sagittal spinal balance parameters. The set of marker-based sagittal spinal balance parameters comprises LL, TK, sagittal vertical axis (SVA), spino-sacral angle (SSA), spine inclination (SI). The data obtained using motion capture will be used to estimate spinal load using musculoskeletal modeling.
Change in Sagittal Spinal Balance assessed using EOS | At baseline and at one-year follow-up
  Sagittal spinal balance parameters from EOS radiological images are calculated semi-automatically using the sterEOS software provided by the EOS company. This workflow allows the calculation of four sagittal spinal balance parameters: SVA, SSA, LL and TK. LL is calculated as the angle between the tangents on the superior L1 and inferior L5 vertebral endplates. TK is calculated as the angle between the tangents on the superior T4 and inferior T12 vertebral endplates. SVA is measured as the horizontal distance between C7 plumb line and the posterior-superior corner of the S1 vertebra. SSA is defined as the angle between the line connecting the center of the C7 vertebra to the center of the S1 endplate and the line parallel to the superior S1 endplate.
Change in Muscle fatigue assessed using electromyography (EMG) | At baseline and at one-year follow-up
  Muscle fatigue will be assessed as the decrease in median EMG frequency.
Change in Muscle fatigue assessed by fatigue exercise duration | At baseline and at one-year follow-up
  The fatigue exercise duration will be measured using a stopwatch. Time is stopped from the point where the patients starts the exercise by no longer supporting the torso with their hands until the termination of the exercise by supporting the torso.
Change in Radiological parameter: Muscle atrophy | At baseline and at one-year follow-up
  The measurement of muscle atrophy allows quantifying abdominal and paraspinal muscle degeneration. The analysis will be performed using ImageJ image analysis software (Version 1.52t, National Institutes of Health, Bethesda, Maryland).
Change in Radiological parameter: Fatty infiltration | At baseline and at one-year follow-up
  The measurement of fatty infiltration allows quantifying abdominal and paraspinal muscle degeneration. The analysis will be performed using ImageJ image analysis software (Version 1.52t, National Institutes of Health, Bethesda, Maryland).
Change in Radiological parameter: Muscle cross-sectional area (CSA) | At baseline and at one-year follow-up
  For L1 to L5, the cross-sectional area (CSA) of the abdominal and paraspinal muscles on each side will be measured, including the multifidus and the erector spinae (longissimus and iliocostalis) muscles, and the CSA of the vertebral body. The relative CSA (rCSA) will be defined as the ratio between muscle CSA and vertebral body CSA and calculated for each level and side. The CSA of lean muscle in the region of interest will be defined as LeanCSA and measured on each side. The ratio of LeanCSA to the paraspinal muscle CSA will be defined as functional CSA (LeanCSA/CSA), represented as % muscle CSA and calculated for each level and side. Overall CSA, rCSA and LeanCSA will be computed as average CSA (aCSA), average rCSA (arCSA) and average LeanCSA (aLeanCSA) across all levels considering the muscle as a single unit for each side.
Change in Radiological parameter: Stenosis severity | At baseline and at one-year follow-up
  Stenosis severity will be classified according to Schizas (Grade A stenosis is the mildest, with abundant cerebrospinal fluid inside the dural sac. In grade B stenosis, the rootlets occupy the whole of the dural sac, but they can still be individualized. In grade C, no rootlets can be recognized but epidural fat can be visualized posteriorly. In grade D, in addition to no rootlets being recognizable, there is no epidural fat posteriorly).
Change in Radiological parameter: Segmental instability | At baseline and at one-year follow-up
  Segmental instability will be determined as a relative shift in anteroposterior position of two adjacent segments between the upright standing radiograph and the lying MRI of more than 3mm.

OTHER OUTCOMES:
Change in Quality of life (EQ-5D-5L) | At baseline and at one-year follow-up
  The EQ-5D-5L comprises 5 questions/dimensions (mobility, self-care, usual activities, pain, depression) with Likert-scale response and a visual analogue scale where patients are asked to rate their overall health from 0 (the worst health imaginable) to 100 (the best health imaginable). Each dimension allows to choose five levels labelled as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression). Using the EQ-5D-5L, a total of 3125 different health states can be described. The final EQ index is a number between 0 and 1, with 0 indicating the poorest possible health (a state as bad as being dead) and 1 indicating the best possible health.
Change in Swiss spinal stenosis score | At baseline and at one-year follow-up
  The Swiss Spinal Stenosis Questionnaire is a self-report outcome questionnaire for patients with LSS and assesses the intensity of symptoms, physical function, and patient satisfaction following treatment.
Change in Tampa scale of kinesiophobia | At baseline and at one-year follow-up
  The Tampa scale is a 17-item self-report questionnaire based on the assessment of fear of exercise, fear of physical activity, and fear avoidance. It consists of two subscales. While activity avoidance revolves around the reflection of activities that may increase pain or cause injury, somatic focus investigates the reflection of beliefs and underlying serious conditions.
Change in Core Outcome Measures Index for the back (COMI back) | At baseline and at one-year follow-up
  The COMI is a validated 11-item self-report questionnaire for assessing the main outcomes of importance to patients back problems.
Change in Upper body motion (inertial sensor data) | At baseline and at one-year follow-up
  During all tasks, inertial sensor data will be collected. Inertial sensors (Blue Trident IMU, Vicon, Oxford, UK) will be placed on the subjects' femora, thoracic and lumbar spine and on the sternum. Accelerations and angular velocity will be captured for all movement assessments.
Change in Manual testing for muscle strength | At baseline and at one-year follow-up
  Selected muscles of the legs will be assessed according to Janda's M5/5 levels of strength. In a sitting position: Hip flexion / M. iliopsoas (L2), Knee extension/ M. quadriceps femoris (L3). In a supine lying position: Foot extension (lift up) / M. tibialis anterior (L4), Lifting the big toe/ M extensor hallucis longus (L5). Foot extension (push down)/ M. gastrocnemius (S1).
Change in Physical activity level | first assessment period: 9 days after the baseline measurement on test day 1; second period: 6 months after the spine surgery; third period: for 9 days at the one-year follow-up visit
  Physical activity (PA) level will be assessed using an activity monitor (GENEActiv, Activinsights, Kimbolton, UK) during three periods of time (9 days each).
Change in Back performance scale | At baseline and at one-year follow-up
  The Back performance scale is an assessment consisting of a series of five movement activities that require mobility of the trunk. The activities (sock test, pick-up test, roll-up test, fingertip-to-floor test, and lift test) all require sagittal-plane mobility and are scored from 0 (can easily do) to 3 (hard/limited to do.

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Netzer, PD Dr. med., Principal Investigator — Department of Spine Surgery, University Hospital Basel
Locations (1):
- Department of Spine Surgery, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Koch D, Nuesch C, Ignasiak D, Aghlmandi S, Caimi A, Perrot G, Prufer F, Harder D, Santini F, Scharen S, Ferguson S, Mundermann A, Netzer C. The role of muscle degeneration and spinal balance in the pathophysiology of lumbar spinal stenosis: Study protocol of a translational approach combining in vivo biomechanical experiments with clinical and radiological parameters. PLoS One. 2023 Oct 27;18(10):e0293435. doi: 10.1371/journal.pone.0293435. eCollection 2023. PMID 37889898